CLINICAL TRIAL: NCT00426790
Title: Open Lung Approach During General Anaesthesia to Prevent Post-Operative Pulmonary Complications
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Università degli Studi dell'Insubria (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1400
Record Dates: First submitted 2007-01-24; First posted 2007-01-25 (Estimated); Last update posted 2007-01-25 (Estimated); Status verified 2007-01

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Positive-Pressure Respiration

INTERVENTIONS:
Procedure: Positive end-expiratory pressure

SUMMARY:
The hypothesis of this study is that the "Open lung approach" ( recruitment and PEEP) during general anaesthesia reduces atelectasis formation and improves respiratory function in the immediate post-operative period after major abdominal surgery.

This is a prospective, randomized, controlled clinical-trial,performed in patients undergoing major abdominal surgery, to compare the effects on the post-operative pulmonary complications of two different intraoperative ventilatory strategies during general anaesthesia: 1- Control Group: PEEP 0 cmH2O without recruitment manoeuvre; 2- Treatment Group:recruitment manoeuvre (after intubation and before extubation) and PEEP 10 cmH2O In the post-operative period the following variables will be recorded at the first, third and fifth postoperative day: 1- Gas-exchange in air; 2- Chest X-ray for atelectasis evaluation; 3- signs of pulmonary complication (cough, secretions, dyspnea, thoracic pain)

ELIGIBILITY:
Inclusion Criteria:

* Patients with ASA 1, 2 and 3
* Age higher than 18 years
* Major abdominal surgery
* General anesthesia

Exclusion Criteria:

* COPD with FEV1 lower than 50%
* Ischemic cardiopathy
* Loco-regional anesthesia alone
* Minor abdominal surgery
* Laparoscopic surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pelosi, Professor, Principal Investigator — University of Insubria, Varese, Italy
Locations (1):
- Ospedale di Circolo e Fondazione Macchi, Varese, Varese, Italy